CLINICAL TRIAL: NCT04680858
Title: Impact of Digital Enhanced Telecommunication for Team Communication in Endoscopic Procedures During COVID-19 Pandemic
Brief Title: Impact of Digital Communication Assist Tools in Endoscopic Team Communication During COVID-19
Acronym: EndoCom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Thomas Seufferlein, Head of Mecical clinic 1, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 122020
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Endoscopy; Communication
Keywords: endoscopy; team communication; endoscopic procedure; COVID-19
MeSH Terms: conditions — Communication; COVID-19

STUDY DESIGN:
Intervention Model Description: Two-armed study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Communication (No Intervention): Endoscopic procedures performed by skilled endoscopic team with standard communication (no headset)
- DECT enhanced Communication (Experimental): Endoscopic procedures performed by skilled endoscopic team with enhanced communication tools ( DECT headset)
  Interventions: Other: DECT

INTERVENTIONS:
Other: DECT — Use of a digital enhanced telecommunication headset for team communication
  Arms: DECT enhanced Communication

SUMMARY:
Team work is highly challenged by the COVID-19 pandemic. Necessary protective equipment as FFP-mask and face shields impair communication significantly.Objective of the study is to evalaute the impact of digital enhanced telecommunication in endoscopic procedures.

DETAILED DESCRIPTION:
Optimal communication is crucial for team work in high class endoscopy. Team work is highly challenged by the COVID-19 pandemic. Necessary protective equipment as FFP-mask and face shields impair communication significantly. Digital enhanced approaches to maintain team communication during endoscopic procedures are mandatory not only in actual circumstances.

Materials and methods:A prospective, two-armed interventional study will be performed at an endoscopy unit at a tertiary center. 200 endoscopic examinations (EGD, colonoscopy, EUS, ERCP) were randomly assigned (1:1) to a group that was performed with DECT equipped endoscopy team or with standard communication. All examinations were performed under protective equipment. Primary outcome was rate of communication associated adverse events. Secondary outcomes included team subjectively perceived comfort with DECT enhanced communication during endoscopic work, duration of examinations, SAE.

ELIGIBILITY:
Inclusion Criteria:

* Member of staff of the endoscopic team (Doctor, nurse)

Exclusion Criteria:

* Deafness
* significantly impaired hearing

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Communication associated adverse events | From start to stop of endoscopic procedure
  Adverse events arising from impaired communication by COVID-19 protection equipment

SECONDARY OUTCOMES:
Severe adverse events | From start to stop of endoscopic procedure
  Severe adverse evatent, not arising from from impaired communication by COVID-19 protection equipment
Subjective Comfort of DECT communication | From start to stop of endoscopic procedure
  Subjectiveley perceived level of comfort using DECT communication during endoscopic procedures rated by numeric rating scale (1-6)
Endoscopic time | From start to stop of endoscopic procedure
  Duration of performed endoscopic procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No